CLINICAL TRIAL: NCT05197465
Title: Persistent Opioid Consumption After Major Abdominal Surgery and Its Determinants: A Prospective Cohort Study
Brief Title: Persistent Opioid Consumption After Major Abdominal Surgery and Its Determinants
Acronym: POCAS
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 21.314
Record Dates: First submitted 2022-01-05; First posted 2022-01-19 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Major Abdominal Surgery; Chronic Pain; Opioid Use
MeSH Terms: conditions — Chronic Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing major abdominal surgery: The investigators aim to conduct a prospective observational, cohort study including all patients undergoing a major open abdominal surgery.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Participants will complete pain and quality of life questionnaires. Opioid consumption will also be assessed using validated questionnaires.

SUMMARY:
The opioid crisis is a growing problem around the world, with prescription opioids being a major contributor to this crisis. They can be prescribed in different chronic and acute settings, such as surgery. This is therefore an event which may mark a first exposure to opioids in many opioid-naive patients and be associated with subsequent long-term use. This long-term persistent opioid consumption (POC) after surgery may be due, among other things, to chronic postsurgical pain (CPSP). Many risk factors have been identified in the development of chronic pain. Some are related to the surgery while others are related to patient characteristics. Of these, preoperative opioid use, pre-existing pain, and psychological history are major factors that increase the risk of POC or CPSP.

The population having undergone major abdominal surgery remains poorly represented in studies of postoperative POC. It can be reasonable to think that these patients may have a similar high risk of CPSP and POC as other surgical patients. The potential harmful effects of POC and CPSP may limit the recovery of these patients and impair their quality of life (QoL).

The risk factors for CPSP are important to consider when considering POC. While psychological factors related to pain have been shown to be associated with postoperative pain and analgesic use, the association between unrelieved postoperative pain and POC may have been underestimated. Regional anesthesia is frequently used in major abdominal surgery to reduce the risk of acute and chronic postoperative pain. However, data regarding CPSP specifically after major abdominal surgery are lacking, and the role of neuraxial analgesia on its prevention and on postoperative opioid use is unclear.

Since little is known about the prevalence of POC after major abdominal surgery and its determinants, the investigators propose to conduct a major abdominal surgery cohort study by examining POC and CPSP using information reported by patients.

DETAILED DESCRIPTION:
Objectives

Primary objective: estimate the prevalence of POC 3 months after major abdominal surgery, describe its distribution in both opioid-naive and chronic opioid users and across different types of abdominal surgery, and estimate its association with persistent pain and quality of life.

Secondary objective: estimate the effects of individual potential risk factors on POC after major abdominal surgery.

Tertiary exploratory objective: evaluate the effect of neuraxial analgesia on POC.

Exploratory objectives: describe distribution of opioid misuse among patients with POC and the opioid consumption trajectory among preoperative chronic opioid users.

The hypotheses of the study are that:

1. POC will be high after abdominal surgeries (close to what has been reported in thoracic surgeries and pancreatectomies) and will be associated with a higher prevalence of persistent pain and lower quality of life,
2. Certain surgical and individual risk factors are determinants of POC,
3. The reduction of acute pain with neuraxial analgesia will help reduce the prevalence of postoperative POC.
4. Opioid misuse will be rare among patients with POC and most preoperative chronic opioid users with POC will not have decreased their consumption.

Design of the study: multicenter, prospective, cohort study. After obtaining consent, consecutive adult patients undergoing major open abdominal surgery will be included over a 6-month period.

Before surgery, data on planned surgery, demographics, socio-economic status, surgical and medical history, including information on preoperative opioid use and preoperative pain will be collected. For chronic opioid users, information about the reasons for opioid consumption will be recorded. Presence of co-morbidities, frailty, anxiety or depressive symptoms, catastrophizing tendency, and quality of life will be assessed using validated questionnaires.

During the hospitalization associated with the index surgery, the following data will be collected: type of anesthesia, administration of opioids or any other analgesic medication, care required following the intervention, quality of pain control, dosage of opioid consumption and presence of an opioid prescription upon discharge from hospital. The need to perform any other surgery during index hospitalization and the use of the pain transition service will be noted.

Patients will be contacted by phone three months after surgery. To quantify opioid use, a Timeline Follow Back questionnaire will be used. This questionnaire will include questions regarding opioids used, dose, frequency of use, mode of administration, reason for use, and presence of other sources of opioids, if applicable (family, unused opioids from old prescriptions). For preoperative opioid users, changes in opioid consumption will be assessed. Pharmacy-reported information regarding served opioid will be collected. The presence of complications related to opioid consumption as well as the risk of misuse will be assessed by using the Opioid Compliance Checklist. Information on hospitalizations associated with opioid-related events and on care level trajectory for up to three months after surgery will be recorded. Postoperative pain and quality of life will be assessed using validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing major open abdominal surgery during the study period (6 months)
* Patients suffering from chronic pain or using opioids may be included since they are at risk of developing CPSP or POC

Exclusion Criteria:

* Patients who have already participated in the study will be excluded as well as patients who will undergo a second surgery after discharge from hospital and before the 90-day deadline for the primary endpoint.
* Patients undergoing appendectomies, inguinal hernia repair and abdominal wall hernia repair other than incisional hernias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators aim to conduct a prospective cohort study. This study will take place at the Centre Hospitalier de l'Université de Montréal (CHUM) and CIUSSS de l'Est-de-l'Île-de-Montréal (Maisonneuve-Rosemont Hospital)
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2022-02-13 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Patient-reported opioid use | 3 months after surgery
  Any consumption of opioids as declared by patients during the 7 days prior to the 3-month interview

SECONDARY OUTCOMES:
Presence of chronic pain and its assessment by BPI | 3 months after surgery
  Presence of persistent pain in the 7 days prior to the interview or worsening of the pain at surgical site for patients who had pain at that site prior to surgery. Pain will be assessed using a modified version of the Brief Pain Inventory (BPI)-short questionnaire, which consists of questions regarding presence, duration and location of pain, pain-relief medication usage, pain intensity using Numeral Rating Scale (NRS), treatment effectiveness in percentage of pain relief ranging from 0 to 100% and impact of pain on quality of life also using NRS. NRS ranges from 0 to 10, 10 meaning the worst outcome.
Change in quality of life assessed by SF-12 | 3 months after surgery
  Quality of life will be assessed at baseline and at 3 months following surgery using the Medical Outcomes Study Short Form Survey (SF-12) questionnaire, which results in 2 scores representing physical and mental health. Both mental and physical health scores range from 0 to 100, and a higher score means a better outcome. The results of the SF-12 completed at 3 months following surgery will be compared to the baseline results.

CONTACTS AND LOCATIONS:
Overall Officials: François Martin Carrier, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (2):
- Canada (2):
  - CIUSS-de-l'Est-de-l'Île-de-Montréal (Hôpital Maisonneuve-Rosemont), Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No